CLINICAL TRIAL: NCT06134141
Title: The Outcome of Interventional Cardiac Catheterization In Pediatric Cardiology Unit, Assiut University Heart Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya zidan sayed gomaa, 71515,Assiut, Assiut University
Other Study IDs: CC OUTCOME
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Catheterization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Describe demographic and clinical data of infant and pediatric with cardiac catheterization who admitted to cardiology unit of Assiut university children hospital Asses outcome of cardiac catheterization in pediatric and infant at AUCH

DETAILED DESCRIPTION:
Cardiac catheterization and intervention in pediatric cardiac diseases have evolved significantly in the past 30 years. During the last 10 years, there have been major technological achievements in pediatric interventional cardiology There have also been substantial advancements in cardiac imaging modalities, such as intracardiac echocardiography (ICE), real-time 3-dimensional (3D) transesophageal echocardiography (TEE), cardiac computed tomography (CT) and magnetic resonance imaging (MRI), rotational angiography with 3D roadmap, holography, 3D printing, and Echo-Navigator and Vessel-Navigator systems. As a result of such technological advances, more types of congenital heart diseases (CHDs) can be treated in the cardiac catheter laboratory today than ever before. Therefore, the possibility exists that many surgical procedures will be replaced by catheter-based procedures

The pediatric interventional cardiology community has continued to develop less invasive solutions for congenital heart defects (CHDs) to minimize the need for open heart surgery and optimize overall outcomes. Many CHDs are effectively managed with transcatheter techniques. Atrial and ventricular septal defects, valve stenosis, patent ductus arteriosus, aortic coarctation, pulmonary artery and vein stenosis and arteriovenous malformations are some examples, routinely treated with catheterization in the pediatric population For most such interventions, these efforts lead to more highly acceptable outcomes and lower complication rates than the alternatives of surgery or no intervention

ELIGIBILITY:
Inclusion Criteria:

children aged 1 month to 18 years old that underwent cardiac catheterization for congenital heart disease management.

-

Exclusion Criteria:

1-Neonate aged less than 1 month and adult >16 years old 2-Patients with chronic renal and hepatic disease could affect results

-

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children aged 1 month to 18 years old that underwent cardiac catheterization for congenital heart disease management.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-17 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
procedure time [ Time Frame: duration of the cardiac catheterization procedure (1-4 hours depending on complexity of case) ] | Baseline
  duration of the cardiac catheterization procedure (1-4 hours depending on complexity of case|)

REFERENCES:
- [Background] Crystal MA, Ing FF. Pediatric interventional cardiology: 2009. Curr Opin Pediatr. 2010 Oct;22(5):567-72. doi: 10.1097/MOP.0b013e32833e1328. PMID 20733492
- [Background] Moustafa GA, Kolokythas A, Charitakis K, Avgerinos DV. Therapeutic Utilities of Pediatric Cardiac Catheterization. Curr Cardiol Rev. 2016;12(4):258-269. doi: 10.2174/1573403x12666160301121253. PMID 26926291
- [Background] Backes CH, Cheatham SL, Deyo GM, Leopold S, Ball MK, Smith CV, Garg V, Holzer RJ, Cheatham JP, Berman DP. Percutaneous Patent Ductus Arteriosus (PDA) Closure in Very Preterm Infants: Feasibility and Complications. J Am Heart Assoc. 2016 Feb 12;5(2):e002923. doi: 10.1161/JAHA.115.002923. PMID 26873689